CLINICAL TRIAL: NCT04781140
Title: A Phase 4, Randomized, Double-Blind, Multicenter, Placebo-Controlled, Parallel-Group Study of the Efficacy and Safety of SPN-812 in Preschool-Age Children (4 to 5 Years Old) With Attention-Deficit/Hyperactivity Disorder (ADHD)
Brief Title: Evaluation of SPN-812 (Viloxazine Extended-release Capsule) in Preschool-age Children With ADHD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 812P401
Record Dates: First submitted 2021-02-26; First posted 2021-03-04 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Attention-Deficit/Hyperactivity Disorder
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo, qd
  Interventions: Drug: Placebo
- SPN-812 (Experimental): SPN-812, qd
  Interventions: Drug: 100mg SPN-812

INTERVENTIONS:
Drug: 100mg SPN-812 — 100mg SPN-812 will be administered once daily and compared to Placebo
  Other Names: SPN-812
  Arms: SPN-812
Drug: Placebo — Placebo will be administered once daily
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of SPN-812 (viloxazine extended release) in children 4 to 5 years of age with ADHD.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multicenter, 2-arm (1:1), parallel-group, efficacy and safety/tolerability fixed-dose study of SPN-812 in preschool-age children (4 to 5 years old) with ADHD. Participants will be screened for eligibility for up to 4 weeks. Eligible participants will be treated with study medication for 6 weeks. The total duration of the study is up to 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Is male or female 4 years 0 months of age to less than or equal to 5 years 9 months of age at Visit 1 (Screening) and considered medically healthy.
2. Subject's parent(s) or legal guardian(s)/representative(s) is (are) willing and able to provide written informed consent before completing any study related procedures.
3. Has a primary diagnosis of ADHD according to DSM-IV-TR criteria and confirmed with the Kiddie Schedule for Affective Disorders and Schizophrenia - Present and Lifetime Version (K-SADS-PL).
4. Has an ADHD-RS-IV-P Total Score of ≥ 28 (males) or ≥ 24 (females) at Visit 1 (Screening) and at Visit 2 (Baseline).
5. Has a CGI-S score of ≥ 4 (moderate or worse) at Visit 1 (Screening) and at Visit 2 (Baseline).
6. Has undergone an adequate course of non-pharmacologic treatment or is having symptoms severe enough to warrant pharmacologic treatment without prior non-pharmacologic treatment.
7. Is participating in a structured group activity (e.g., preschool, kindergarten, sports, Sunday school, summer camp or childcare program) at least 2 days a week during study so as to assess symptoms and impairment in a setting outside the home.
8. Has not initiated any behavioral intervention/therapy within 30 days of Visit 1 (Screening) and does not plan to initiate any new or discontinue any ongoing behavioral intervention/therapy during the study (e.g., subject is eligible if behavioral intervention/therapy is initiated 30 or more days prior to Visit 1 [Screening] and continues with a similar duration/frequency throughout their study).
9. Subjects who are on ADHD medication at Visit 1 (Screening), but whose ADHD symptoms are not well controlled on current ADHD medication (e.g., meets Inclusion Criterion #4), meet all other inclusion/exclusion criteria, and discontinues ADHD medication at least 7 days prior to the day of Visit 2 (Baseline) are eligible to participate.
10. Has no current condition in the opinion of the Investigator that could confound efficacy assessments, safety assessments or increase participant risk.
11. Has lived with the same parent(s) or legal guardian(s) or has lived under a shared living arrangement (e.g., joint legal custody) for greater than or equal to 6 months prior to Visit 1 (Screening).
12. Has a body weight ≥5th percentile for age and sex at Visit 1 (Screening) and Visit 2 (Baseline).

Exclusion Criteria:

1. Has a diagnosis at Screening (per K-SADS-PL) of another psychiatric disorder that is considered to be the primary diagnosis rather than ADHD or has a comorbid psychiatric disorder secondary to ADHD that, in the opinion of the investigator (after consulting medical monitor), will likely interfere with study treatment adherence and/or impact study results.
2. Has a current diagnosis of a major neurological disorder. The eligibility of those who have seizures, a history of seizure-like events (e.g., syncope, myoclonus, severe muscle spasms), a family history of seizure disorder (immediate family, i.e., sibling, parent), and/or febrile seizures will be assessed on a case-by-case basis after consulting the medical monitor.
3. History of Bipolar Disorder diagnosed in a first degree relative.
4. Has global development delay or intellectual disability by medical history.
5. Has a current diagnosis of a significant (per Investigator's evaluation and/or judgement) systemic disease.
6. Has body mass index > 95th percentile for the subject's age and sex at Visit 1 (Screening) or Visit 2 (Baseline).
7. Has a mean resting systolic and diastolic blood pressure* that are both >95th percentile for age sex, and height and has a mean resting pulse rate* that is >95th percentile for age and sex (males: >117 bpm; females: >122 bpm) at Visit 1 (Screening) or Visit 2 (Baseline). * Note: The mean of three measurements while seated.
8. Has a clinically significant electrocardiogram finding(s) at Visit 1 (Screening).
9. Is currently taking SPN-812 for ADHD, has previously taken SPN-812 for ADHD, but discontinued due to a lack of efficacy or adverse reactions, or has history of allergic reaction, hypersensitivity or intolerance to viloxazine.
10. Has an allergy to or cannot swallow pudding and applesauce and cannot swallow intact capsule whole.
11. Has any food allergy, intolerance, restriction or special diet that, in the opinion of the Investigator, could contraindicate the subject's participation in the study.
12. Has received any investigational drug within the longer of 30 days or 5 half-lives prior to Visit 2 (e.g., first dose of study medication).
13. Has a positive urine drug test at Visit 1 (Screening). A positive test for amphetamines is allowed for subjects receiving a stimulant ADHD medication at Screening. The subject will be required to discontinue the stimulant for the duration of the study, beginning at least 7 days prior to Visit 2 (Baseline).
14. Is using of prohibited concomitant medications including known CYP1A2 substrates (e.g., theophylline, melatonin) during the Screening Period or (anticipated) for the duration of the study.
15. Any reason that, in the opinion of the Investigator, would prevent the subject from participating in the study.
16. Has suicidal ideation ("Yes" indicated on C-SSRS question 4 or 5) or suicidal behavior ("Yes" indicated on C-SSRS for any suicidal behavior) within 6 months prior to or the day of Visit 1 (Screening) or has attempted suicide ("Yes" indicated on C-SSRS for lifetime).

Ages: 48 Months to 69 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 286 (Estimated)
Dates: Start 2024-03-19 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Attention-Deficit/Hyperactivity Disorder Rating Scale, 4th Edition, Preschool Version (ADHD-RS-IV-P) Total Score at End of Study (Week 6) | Baseline and Week 6
  The Attention-Deficit/Hyperactivity Disorder Rating Scale, 4th Edition, Preschool Version (ADHD-RS-IV-P) consists of 18 items that correspond directly to the DSM-IV-TR criteria for ADHD. The scale is subdivided into two subscales: inattention ("IA", 9 items) and hyperactivity-impulsivity ("H/I", 9 items).The clinician rates the frequency and severity of each symptom on a 4-point Likert-type scale, where 0 = Never or rarely, 1 = Sometimes, 2 = Often, and 3 = Very often. The sum of the ratings of all 18 items yields the raw Total score (range: 0-54; the higher the Total score, the more severe the ADHD symptoms). Post-baseline raw Total scores are converted to a change from baseline Total score. A lower change from baseline ADHD-RS-IV-P Total Score (<0) represents a better outcome.

SECONDARY OUTCOMES:
Change from Baseline in the Clinical Global Impression of Severity (CGI-S) Score at End of Study (Week 6) | Baseline and Week 6
  The Clinical Global Impression of Severity (CGI-S) is a single item clinician-rated assessment of the severity of subject's condition (ADHD symptoms) in relation to the clinician's total experience with patients with ADHD. The CGI-S is evaluated on a 7-point scale with 1 = Normal, not at all ill, asymptomatic, 2 = Borderline Ill, 3 = Mildly Ill, 4 = Moderately Ill, 5 = Markedly Ill, 6 = Severely Ill, and 7 = Among the most extremely ill patients (the higher the score, the more severe the overall ADHD symptoms). Post-baseline (raw) CGI-S scores are converted to a change from baseline score. A lower change from baseline CGI-S score (<0) represents a better outcome.
Clinical Global Impression of Change (CGI-C) Score at End of Study (Week 6) | Week 6
  The Clinical Global Impression of Change (CGI-C) is a single item clinician-rated assessment of how much the subject's condition (ADHD) has improved, worsened or has not changed relative to his/her baseline state prior to the beginning of treatment. The CGI-C is rated on a 7-point scale from 1 to 7, where 1 = "very much improved", 2 = "much improved", 3 = "minimally improved", 4 = "no change", 5 = "minimally worse", 6 = "much worse", and 7 = "very much worse". A CGI-C score <4 represents a better outcome.
Change from Baseline in Attention-Deficit/Hyperactivity Disorder Rating Scale, 4th Edition, Preschool Version (ADHD-RS-IV-P) Hyperactivity/Impulsivity Subscale Score at End of Study (Week 6) | Baseline and Week 6
  The Attention-Deficit/Hyperactivity Disorder Rating Scale, 4th Edition, Preschool Version (ADHD-RS-IV-P) consists of 18 items that correspond directly to the DSM-IV-TR criteria for ADHD. The scale is subdivided into two subscales: inattention ("IA", 9 items) and hyperactivity-impulsivity ("H/I" 9 items).The clinician rates the frequency and severity of each symptom on a 4-point Likert-type scale, where 0 = Never or rarely, 1 = Sometimes, 2 = Often, and 3 = Very often. The sum of the nine H/I items yields the raw H/I subscale score (range: 0-27; the higher the H/I subscale score, the more severe the H/I symptoms). Post-baseline raw H/I subscale scores are converted to a change from baseline score. A lower change from baseline H/I subscale score (<0) represents a better outcome.
Change from Baseline in Attention-Deficit/Hyperactivity Disorder Rating Scale, 4th Edition, Preschool Version (ADHD-RS-IV-P) Inattention Subscale Score at End of Study (Week 6) | Baseline and Week 6
  The Attention-Deficit/Hyperactivity Disorder Rating Scale, 4th Edition, Preschool Version (ADHD-RS-IV-P) consists of 18 items that correspond directly to the DSM-IV-TR criteria for ADHD. The scale is subdivided into two subscales: inattention ("IA", 9 items) and hyperactivity-impulsivity ("H/I" 9 items).The clinician rates the frequency and severity of each symptom on a 4-point Likert-type scale, where 0 = Never or rarely, 1 = Sometimes, 2 = Often, and 3 = Very often. The sum of the nine IA items yields the raw IA subscale score (range: 0-27; the higher the IA subscale score, the more severe the IA symptoms). Post-baseline raw IA subscale scores are converted to a change from baseline score. A lower change from baseline IA subscale score (<0) represents a better outcome.
Clinical Global Impression of Severity (CGI-S) Responder Rate (percentage of subjects with CGI-S score of 1 or 2) at End of Study (Week 6) | Baseline and Week 6
  The Clinical Global Impression of Severity (CGI-S) is a single item clinician-rated assessment of the severity of subject's condition (ADHD symptoms) in relation to the clinician's total experience with patients with ADHD. The CGI-S is evaluated on a 7-point scale with 1 = Normal, not at all ill, asymptomatic, 2 = Borderline Ill, 3 = Mildly Ill, 4 = Moderately Ill, 5 = Markedly Ill, 6 = Severely Ill, and 7 = Among the most extremely ill patients. The responder rate (percent) is calculated by dividing "the number of 'responders' (m)" by "the number of subjects analyzed at the respective Visit/Week (n)" and multiplying the product by 100. Responder Rate values range from 0 to 100%. A percent >50% represents a greater number of "responders" versus "non-responders".
Clinical Global Impression of Change (CGI-C) Responder Rate (percentage of subjects with CGI-C score of 1 or 2) at End of Study (Week 6) | Week 6
  The Clinical Global Impression of Change (CGI-C) is a single item clinician-rated assessment of how much the subject's condition (ADHD) has improved, worsened or has not changed relative to his/her baseline state prior to the beginning of treatment. The CGI-C is rated on a 7-point scale from 1 to 7, where 1 = "very much improved", 2 = "much improved", 3 = "minimally improved", 4 = "no change", 5 = "minimally worse", 6 = "much worse", and 7 = "very much worse". The responder rate (percent) is calculated by dividing "the number of 'responders' (m)" by "the number of subjects analyzed at the respective Visit/Week (n)" and multiplying the product by 100. Responder Rate values range from 0 to 100%. A percent >50% represents a greater number of "responders" versus "non-responders".
Attention-Deficit/Hyperactivity Disorder Rating Scale, 4th Edition, Preschool Version (ADHD-RS-IV-P) Responder Rate (percentage of subjects with ≥ 50% Reduction in Change from Baseline) at End of Study (Week 6) | Baseline and Week 6
  The Attention-Deficit/Hyperactivity Disorder Rating Scale, 4th Edition, Preschool Version (ADHD-RS-IV-P) consists of 18 items that correspond directly to the DSM-IV-TR criteria for ADHD. The scale is subdivided into two 9 item subscales: inattention and hyperactivity-impulsivity. The clinician rates the frequency and severity of each symptom on a 4-point Likert-type scale; 0 = Never or rarely, 1 = Sometimes, 2 = Often, and 3 = Very often. Sum of 18 ratings yields the Total score (range: 0-54; higher score represents severer symptoms). Percent reduction is calculated for the ADHD-RS-IV-P score: [("Post-baseline"-"Baseline")/"Baseline"] x 100; range: 0 to 100%; a "responder" is a subject with a 50% or greater reduction in change from baseline Total score. Responder rate (percent of responders) is calculated: ["number of 'responders' (m)"/ "number of subjects analyzed" (n)] X 100; range: 0 to 100%. A Responder Rate greater than 50%, represents more "responders" versus "nonresponders".

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Rubin, MD, MBA, Study Director — Supernus Pharmaceuticals, Inc.
Locations (47):
- United States (47):
  - The Center for Clinical Trials, Inc., Saraland, Alabama
  - Preferred Research Partners, Inc., Little Rock, Arkansas
  - Advanced Research Center (ARC), Inc., Anaheim, California
  - Sun Valley Research Center, Imperial, California
  - Alliance Research, Long Beach, California
  - IMMUNOe Research Centers, Centennial, Colorado
  - Luna Research Center, Coral Gables, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Avantis Clinical Research LLC, Miami, Florida
  - Hope Research Network, LLC., Miami, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - APG Research LLC, Orlando, Florida
  - D&H Tamarac Research Center, Tamarac, Florida
  - Pediatric Neurology and Epilepsy Specialists, Winter Park, Florida
  - Advanced Discovery Research LLC, Atlanta, Georgia
  - Clinical Integrative Research Center of Atlanta, Atlanta, Georgia
  - CenExcel iResearch, LLC, Decatur, Georgia
  - CenExel iResearch, LLC., Savannah, Georgia
  - Qualmedica Research, LLC., Evansville, Indiana
  - Kentucky Pediatric/Adult Research, Bardstown, Kentucky
  - Qualmedica Research, LLC., Owensboro, Kentucky
  - DelRicht Research (Touro Medical Center), New Orleans, Louisiana
  - DelRicht Research, Prairieville, Louisiana
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Neurobehavioral Medicine Group, Bloomfield Hills, Michigan
  - Precise Research Centers, Flowood, Mississippi
  - Clinical Research of Southern Nevada, LLC., Las Vegas, Nevada
  - Med Clinical Research, Irvington, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Hospital and Medical Center, Cincinnati, Ohio
  - CincyScience, West Chester, Ohio
  - Cyn3rgy Research, Gresham, Oregon
  - Penn State Health Medical Group - Psychiatry and Behavioral Health, Hershey, Pennsylvania
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Coastal Pediatric Research, Summerville, South Carolina
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Houston Clinical Trials, LLC., Bellaire, Texas
  - Javara, Dallas, Texas
  - AIM Trials, LLC, Plano, Texas
  - Family Psych of The Woodlands, The Woodlands, Texas
  - Clinical Research Partners, LLC, Petersburg, Virginia
  - Virginia Commonwealth University, Virginia Treatment Center for Children, Richmond, Virginia